CLINICAL TRIAL: NCT00100269
Title: A Randomized Control Trial of the Menevit Anti-Oxidant Therapy for the Treatment of Male Infertility
Brief Title: Menevit Study: Menevit Anti-Oxidant Therapy for the Treatment of Male Infertility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repromed (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCHDW002
Record Dates: First submitted 2004-12-27; First posted 2004-12-28 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2005-06

CONDITIONS: Infertility, Male; Oxidative Stress
Keywords: Male infertility; sperm; pregnancy; IVF (in vitro fertilisation); oxidative stress; free radicals; DNA damage
MeSH Terms: conditions — Infertility, Male

INTERVENTIONS:
Drug: Menevit anti-oxidant

SUMMARY:
Oxidative stress related damage to sperm is believed to be a major cause of male infertility. The object of the Menevit study is to investigate the role of a novel anti-oxidant preparation (Menevit) on sperm function, embryo quality and pregnancy rates in an in vitro fertilization (IVF) setting.

DETAILED DESCRIPTION:
Men will be screened for oxidative stress (free radical) related damage to their sperm. This will include screening for lipid peroxidation of sperm using the LPO-586 assay, HOST test and for sperm DNA fragmentation using the Tunel technique. Those men found to have free radical related damage will be enrolled in a randomized control trial in which they will receive either the Menevit anti-oxidant or placebo (in a 2:1 randomization ratio respectively). The Menevit anti-oxidant is a capsule containing several different anti-oxidants, taken orally once per day. The placebo is identical in appearance and taste. After 3 months of Menevit/placebo the female partners of these men will undergo an IVF oocyte retrieval operation and embryo transfer. Pregnancy rates and embryo quality will be compared between groups. Changes in semen characteristics (count, motility, morphology, membrane integrity) and lipid peroxidation (LPO-586) plus sperm DNA fragmentation (Tunel assay) will be assessed at trial entry, 6 weeks and 3 months. Comparisons between the patients embryo quality in the IVF cycle immediately before and during the Menevit trial will also be compared when possible

ELIGIBILITY:
Inclusion Criteria:

* Evidence of oxidative stress to sperm on LPO-586 assay or poor HOST result or clinical evidence for oxidative stress (heavy smoker, varicocele, poor motility in the abscence of anti-sperm antibodies etc)
* Evidence of significant sperm DNA damage (25% or more DNA fragmentation as assessed by Tunel assay).
* Female partner willing to undergo IVF treatment within 3 months of starting Menevit trial

Exclusion Criteria:

* Female partner 40 years of age or older at trial entry.
* Significantly reduced ovarian reserve in female partner (day 3-5 FSH > 10 iu/L if no prior IVF cycle or less than 5 oocytes on a prior IVF cycle.
* Sperm count below 0.5 million per ml (impossible to conduct all sperm function assays

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-12; Study Completion 2006-03

PRIMARY OUTCOMES:
Embryo quality (morphology score, progression to blastocyst rates, number of embryos available for freezing/transfer per cycle)
Embryo quality is a good measure of pregnancy potential and is also an indicator of sperm DNA integrity, making it the ideal primary endpoint.

SECONDARY OUTCOMES:
sperm DNA fragmentation
sperm count
sperm motility (total motile sperm per ejaculate)
sperm morphology
sperm membrane integrity (as assessed by hypo-osmolar swelling test)
levels of sperm lipid peroxidation (LPO-586 assay)
retrospective comparison of embryo quality between the Menevit IVF cycle and the preceding non-Menevit IVF cycle.
miscarriage rate (clinical and biochemical)
clinical pregnancy rates (number of fetal hearts seen on first trimester scan)
adverse side effects

CONTACTS AND LOCATIONS:
Overall Officials: Kelton P Tremellen, MB BS (Hons) PhD, Principal Investigator — Repromed, University of Adelaide
Locations (1):
- Repromed, Adelaide, South Australia, Australia

REFERENCES:
- [Background] Aitken RJ, Baker MA. Oxidative stress and male reproductive biology. Reprod Fertil Dev. 2004;16(5):581-8. doi: 10.10371/RD03089. PMID 15367373
- [Background] Aitken RJ, Gordon E, Harkiss D, Twigg JP, Milne P, Jennings Z, Irvine DS. Relative impact of oxidative stress on the functional competence and genomic integrity of human spermatozoa. Biol Reprod. 1998 Nov;59(5):1037-46. doi: 10.1095/biolreprod59.5.1037. PMID 9780307
- [Background] Benchaib M, Braun V, Lornage J, Hadj S, Salle B, Lejeune H, Guerin JF. Sperm DNA fragmentation decreases the pregnancy rate in an assisted reproductive technique. Hum Reprod. 2003 May;18(5):1023-8. doi: 10.1093/humrep/deg228. PMID 12721180
- [Background] Henkel R, Hajimohammad M, Stalf T, Hoogendijk C, Mehnert C, Menkveld R, Gips H, Schill WB, Kruger TF. Influence of deoxyribonucleic acid damage on fertilization and pregnancy. Fertil Steril. 2004 Apr;81(4):965-72. doi: 10.1016/j.fertnstert.2003.09.044. PMID 15066449
- [Background] Carrell DT, Liu L, Peterson CM, Jones KP, Hatasaka HH, Erickson L, Campbell B. Sperm DNA fragmentation is increased in couples with unexplained recurrent pregnancy loss. Arch Androl. 2003 Jan-Feb;49(1):49-55. doi: 10.1080/01485010290099390. PMID 12647778
- [Background] Agarwal A, Nallella KP, Allamaneni SS, Said TM. Role of antioxidants in treatment of male infertility: an overview of the literature. Reprod Biomed Online. 2004 Jun;8(6):616-27. doi: 10.1016/s1472-6483(10)61641-0. PMID 15169573
- [Background] Gomez E, Irvine DS, Aitken RJ. Evaluation of a spectrophotometric assay for the measurement of malondialdehyde and 4-hydroxyalkenals in human spermatozoa: relationships with semen quality and sperm function. Int J Androl. 1998 Apr;21(2):81-94. doi: 10.1046/j.1365-2605.1998.00106.x. PMID 9675617